CLINICAL TRIAL: NCT00090012
Title: The Comparison of Efficacy and Safety of Continuing Olanzapine to Switching to Quetiapine in Overweight or Obese Patients With Schizophrenia and Schizoaffective Disorder
Brief Title: Comparison of Continuing Olanzapine to Switching to Quetiapine in Overweight or Obese Patients With Schizophrenia and Schizoaffective Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8894; F1D-US-HGLR
Record Dates: First submitted 2004-08-18; First posted 2004-08-23 (Estimated); Last update posted 2007-11-06 (Estimated); Status verified 2007-11

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Olanzapine; Quetiapine Fumarate

INTERVENTIONS:
Drug: Olanzapine
Drug: Quetiapine

SUMMARY:
The purposes of this study are to determine:

* The effectiveness of olanzapine as compared to quetiapine in treating and preventing the recurrence of a variety of symptoms of schizophrenia and schizoaffective disorder in patients who are obese or overweight.
* The safety of olanzapine as compared to quetiapine.

ELIGIBILITY:
Inclusion Criteria:

* You must be 18-75 years of age and be diagnosed with schizophrenia or schizoaffective disorder
* You must be able to visit the doctor's office thirteen (13) times over a twenty-six (26) week period

Exclusion Criteria:

* You are a woman and are pregnant or breastfeeding
* You have an acute or unstable medical illness, such as heart, liver, or kidney disease, or you have a seizure disorder. (Note: If you are uncertain about a particular condition, please discuss it with your physician.)
* You have a history of allergic reaction or intolerance to olanzapine or quetiapine

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340
Dates: Start 2004-07; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to assess the treatment difference in time to relapse while on olanzapine 7.5-20 mg/day versus quetiapine 300-800 mg/day in the treatment of obese or overweight patients
with schizophrenia or schizoaffective disorder. Relapse is defined as the occurrence of at least one of the following three conditions:
Hospitalization for psychiatric reasons after Visit 2, or
20% worsening on the Positive and Negative Syndrome Sale (PANSS) Total and an increase in level of care, as compared to Visit 2, or
20% worsening on the PANSS Total compared to Visit 2 and worsening of CGI-S by at least one level compared to Visit 2 and CGI-S level of at least 4 (moderately ill).

SECONDARY OUTCOMES:
To assess within and between group changes in metabolic parameters including fasting glucose, hemoglobin Alc, lipids, and insulin
To assess within and between group changes in weight, waist circumference, BMI, appetite, and prevalence of patients meeting criteria for the metabolic syndrome
To assess within and between group changes in metabolic parameters (fasting glucose and lipids, and hemoglobin A1c) in a sub-group of patients with pre-existing diabetes prior to study entry
To assess the effect of olanzapine versus quetiapine on time to discontinuation for any reason, or lack of efficacy or worsening of psychiatric syndromes
To assess the efficacy of olanzapine versus quetiapine in improving psychopathology of schizophrenia as measured by a mean change from baseline on the PANSS and the Clinical Global Impression-Severity (CGI-S)
Scale as well as by absolute score of CGI-I (Improvement Scale)
To assess the efficacy of olanzapine versus quetiapine in improving depressive symptoms as measured by a mean change from baseline on the montgomery-Asberg Depression Rating Scale (MADRS)
To assess the efficacy of olanzapine versus quetiapine in improving patients' general well being and overall level of functioning as measured by the Short Form 36 Health Survey (SF-36), the Patient Global Impression (PGI)Scale,
and the Global Assessment of Functioning (GAF) Scale
To assess patients' opinions on the treatment with olanzapine versus quetiapine as measured by the Drug Attitude Inventory (DAI-10) Scale
To compare the utilization of medical resources between patients treated with olanzapine or quetiapine
To assess the safety of olanzapine and quetiapine as determined by:
Treatment-emergent adverse events
Vital signs and fasting laboratory analytes
Extrapyramidal symptoms as measured by the Modified Simpson-Angus Scale, the Barnes Akathisia Rating Scale, and the Abnormal Involuntary Movement Scale (AIMS)
A sensitivity analysis will be performed on two randomly chosen subsamples of the overall patient population by analyzing the primary objective respectively

CONTACTS AND LOCATIONS:
Overall Officials: Call1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (25):
- United States (25):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Garden Grove, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Mesa, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Washington D.C., District of Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Granite City, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lafayette, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lake Charles, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Detroit, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashua, New Hampshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Clementon, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kenilworth, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Neptune City, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Princeton, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brooklyn, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Olean, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rochester, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cleveland, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Springfield, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paoli, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Conroe, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Waco, Texas

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com